CLINICAL TRIAL: NCT00356863
Title: The Influence of Increasing Awareness of Cardiac Patients Undergoing Coronary Artery Bypass Grafting (CABG) Surgery to Cardiac Rehabilitation (CR) on Actual Participation Rates and; Patients' Related Barriers to CR Programs Participation
Brief Title: Effect of an Educational Intervention on Cardiac Patients' Participation Rate in Cardiac Rehabilitation Programs
Acronym: MECRIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: The Gertner Institute (Other); Israel National Institute for Health Policy and Health Services Research (Other Government)
Responsible Party: Principal Investigator, Dr. Rachel Dankner, Senior investigator, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SHEBA-05-2374-RD-CTIL
Record Dates: First submitted 2006-07-25; First posted 2006-07-26 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-10

CONDITIONS: Coronary Artery Disease
Keywords: Intervention; Awareness; Cardiac Rehabilitation (CR); Coronary Artery Patients; Coronary Artery Bypass Grafting Surgery (CABG)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Explanation on cardiac rehabilitation (Experimental): Intervention: Increasing awareness to cardiac rehabilitation programs: Patients received a written and oral short explanation on the importance and benefits of cardiac rehabilitation (CR) participation, and information on available programs. They were telephoned 2 weeks after hospital discharge to encourage them to enroll at a cardiac rehabilitation program (CRP). In addition, physicians and nurses at the cardiothoracic units participated in a 1-hour seminar on CR. A recommendation to the general physician to refer the patient to CRP was added to the letter of discharge from hospital.
  Interventions: Behavioral: Increasing awareness to cardiac rehabilitation programs
- Usual care with no intervention (No Intervention): Patients recruited to the study received the usual care without any additional explanation on cardiac rehabilitation, and no effort to increase their awareness or the ward's awareness to cardiac rehabilitation was done.

INTERVENTIONS:
Behavioral: Increasing awareness to cardiac rehabilitation programs — Increasing awareness to cardiac rehabilitation programs: Before coronary artery bypass grafting (CABG) surgery patients received a face-to-face explanation on their right to participate in cardiac rehabilitation programs (CRPs) under the Israeli Basket of Health Services; they were also provided with a brochure on the benefits of CRP participation and the availability of CRPs throughout the country.
  Other Names: Improving participation at cardiac rehabilitation programs
  Arms: Explanation on cardiac rehabilitation

SUMMARY:
The main aim of the study is to determine the effectiveness of an educational intervention designed to increase attendance of coronary artery bypass grafting (CABG) patients at Cardiac Rehabilitation Programs (CRPs) on actual CRP participation rate and; examine patient-related factors (demographic, health, psychosocial, awareness) influencing patients' attendance at CRPs. We hypothesized that the proportion of CABG patients participating in CRPs will increase significantly to 20-30% following the educational intervention employed.

DETAILED DESCRIPTION:
Coronary heart disease (CHD) is a major cause of disability and economic burden in western societies. Ample evidence exists to suggest that participation of these patients in structured Cardiac Rehabilitation Programs (CRPs) is beneficial in terms of improved prognosis and quality of life. Despite inclusion of cardiac rehabilitation (CR) in the Medical Insurance Basket (MIB) as a treatment for patients after an acute myocardial infarction (MI), for those after coronary artery bypass grafting (CABG), and more recently for patients suffering from congestive heart failure, only a small proportion (5%-7.5%) of patients take part in CRPs in Israel. Several factors have been identified as barriers to CRP in Israel, two of which are lack of patients motivation to participate in CRPs stemming, in part, from lack of awareness regarding the importance of CR and its availability and; Lack of motivation of medical staff to refer patients to CR resulting from a unawareness of the importance of CR and its availability across Israel, to name a few. The present study accords with such recommendations, by proposing a simple intervention designed to improve patients' and medical staff's awareness to the importance of CR participation. It is expected that CRP participation will significantly increase to 20-30% following the educational intervention employed.

This intervention will provide the basis for the implementation of an intervention to increase CRP participation in cardiac patients at a national level.

In addition to increasing the proportion of CABG patients attending at CRPs, the study aims to measure the effect of CRP participation on subsequent 1-year health and behavior related outcomes, and 3-year mortality. We expect to find differences in outcome measures between participating patients and those who do not.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Coronary Artery Bypass Grafting with or without valve replacement

Exclusion Criteria:

* Institutionalized patients
* Patients with severe co-morbidities for whom cardiac rehabilitation (CR) is contra-indicated
* Patients who sustained a severe surgical complication preventing them from participating in CR (general stroke with severe disability)
* Patients residing farther than 30 km from a rehabilitation center

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1024 (Actual)
Dates: Start 2004-02; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Dankner, MD MPH, Principal Investigator — The Gertner Institute for Epidemiology and Health Service Research, Sheba Medical Center
Locations (1):
- Sheba Medical Center, the Gertner institute for epidemiology and health service research, Ramat Gan, Israel

REFERENCES:
- [Background] Dankner R, Drory Y, Geulayov G, Ziv A, Novikov I, Zlotnick AY, Moshkovitz Y, Elami A, Schwammenthal E, Goldbourt U. A controlled intervention to increase participation in cardiac rehabilitation. Eur J Prev Cardiol. 2015 Sep;22(9):1121-8. doi: 10.1177/2047487314548815. Epub 2014 Sep 2. PMID 25183694
- [Result] Gendler Y, Geulayov G, Ziv A, Novikov I, Dankner R; Multi-Center Cardiac Rehabilitation Israeli Working Group. [A multicenter intervention study on referral to cardiac rehabilitation after coronary artery bypass graft surgery: a 1-year follow-up of rehabilitation rates among USSR-born and veteran Israeli patients]. Harefuah. 2012 Sep;151(9):511-7, 558, 557. Hebrew. PMID 23367742
- [Result] Dankner R, Geulayov G, Ziv A, Novikov I, Goldbourt U, Drory Y. The effect of an educational intervention on coronary artery bypass graft surgery patients' participation rate in cardiac rehabilitation programs: a controlled health care trial. BMC Cardiovasc Disord. 2011 Oct 8;11:60. doi: 10.1186/1471-2261-11-60. PMID 21982052
- [Derived] Moshkovitz Y, Orenstein L, Olmer L, Laufer K, Ziv A, Dankner R. Emulated Trial for Discharge Prescription of Guideline-Directed Medical Therapy and 15-Year Survival After Coronary Artery Bypass Graft Surgery. Mayo Clin Proc. 2024 May;99(5):766-779. doi: 10.1016/j.mayocp.2023.06.022. Epub 2024 Mar 7. PMID 38456874
- [Derived] Geulayov G, Novikov I, Dankner D, Dankner R. Symptoms of depression and anxiety and 11-year all-cause mortality in men and women undergoing coronary artery bypass graft (CABG) surgery. J Psychosom Res. 2018 Feb;105:106-114. doi: 10.1016/j.jpsychores.2017.11.017. Epub 2017 Dec 1. PMID 29332626
- See also: THE PSYCHOMETRIC PROPERTIES OF THE RUSSIAN VERSION OF THE MACNEW HEART DISEASE HEALTH-RELATED QUALITY OF LIFE SCALE IN PATIENTS UNDERGOING CORONARY ARTERY BYPASS GRAFTING SURGERY — http://bjll.org/index.php/ejpch/article/view/684
- See also: Validation of the Hebrew Version of the MacNew Heart Disease Healthrelated Quality of Life Questionnaire in Patients Undergoing Coronary Artery Bypass Surgery — https://www.omicsonline.org/validation-of-the-hebrew-version-of-the-macnew-heart-disease-healthrelated-quality-of-life-questionnaire-in-patients-undergoing-coronary-artery-bypass-surgery-2155-9880.1000279.php?aid=21660

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All cardiac patients hospitalized in 5 cardiothoracic clinics for coronary artery bypass grafting (CABG) surgery (with or without valve replacement) were offered to participate in the study based on inclusion criteria. Recruitment started on January 2004 and ended on November 2006.
Pre-assignment Details: All first 520 recruited participants from the 5 cardiothoracic units belonged to the control arm of the study and received usual care. The following 504 patients recruited in the 5 cardiothoracic units belonged to the intervention arm and received the educational intervention materials of the study regarding cardiac rehabilitation treatment.
Groups:
- Education (Intervention) Regarding Cardiac Rehabilitation (CR): Cardiac patients were encouraged to participate in cardiac rehabilitation (CR) following coronary artery bypass grafting (CABG) surgery. Medical staff in the operating cardiothoracic units (surgeons and nurses) were encouraged to refer patients to CR.
- No Education (Control) Regarding Cardiac Rehabilitation (CR): Cardiac patients undergoing coronary artery bypass grafting (CABG) surgery receive the usual care without being exposed to the educational intervention. The staff in the cardiothoracic units (surgeons and nurses) did not receive any information about cardiac rehabilitation (CR) and were giving the usual care.
Period: Overall Study
Arm/Group | Education (Intervention) Regarding Cardiac Rehabilitation (CR) | No Education (Control) Regarding Cardiac Rehabilitation (CR)
Started | 504 | 520
Completed | 412 | 445
Not Completed | 92 | 75
Not completed — Death | 16 | 32
Not completed — Lost to Follow-up | 76 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Education (Intervention) Regarding Cardiac Rehabilitation (CR) | No Education (Control) Regarding Cardiac Rehabilitation (CR) | Total
Number analyzed (Participants) | 504 | 520 | 1024
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.644 (9.904) | 66.146 (10.789) | 65.902 (10.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 134 | 244
  Male | 394 | 386 | 780
Region of Enrollment [Number; unit: participants]
  Israel | 504 | 520 | 1024

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Participating in Cardiac Rehabilitation Programs (CRPs)1-year Post Coronary Artery Bypass Grafting (CABG)Surgery in the Intervention and Control Groups
Description: The number of cardiac patients who participated in cardiac rehabilitation programs during the year following coronary artery bypass grafting surgery in the control and the intervention groups.
Time Frame: 1 year
Population: All patients alive at 1-year follow up who gave information on participation in cardiac rehabilitation programs (CRPs) at any time during the year following surgery (and before follow up assessment). This information was obtained via a face-to-face interview or by telephone interview.
Measure: Number; unit: participants
Groups:
- Education (Intervention) on Cardiac Rehabilitation (CR): Cardiac patients were encouraged to participate in cardiac rehabilitation (CR) following coronary artery bypass grafting (CABG) surgery. Medical staff in the operating cardiothoracic units (surgeons and nurses) were encouraged to refer patients to CR.
- No Education (Control) Regarding Cardiac Rehabilitation (CR): Cardiac patients undergoing coronary artery bypass grafting (CABG) surgery receive the usual care without being exposed to the educational intervention. The staff in the cardiothoracic units (surgeons and nurses) did not receive any information about CR and were giving the usual care.
Arm/Group | Education (Intervention) on Cardiac Rehabilitation (CR) | No Education (Control) Regarding Cardiac Rehabilitation (CR)
Number analyzed (Participants) | 450 | 454
participants | 156 | 86

2. Other Pre Specified Outcome: Cardiovascular Morbidity
Description: All hospitalizations which occured during the 1 year follow-up and were due to acute myocardial infarction (International Classification of Disease 9th version (ICD-9) codes 410.), angina pectoris (ICD-9 codes 413.9), stroke/ transient ischemic attack (TIA) (ICD-9 codes 436.), and all surgical procedures which occured during the 1 year follow-up: CABG or coronary catheterizations (ICD-9 codes 36.), endarterectomies (ICD-9 codes 38.0 and 39.0).
Time Frame: 1 year
Population: All patients who were exposed to the educational intervention at baseline and who were contacted a year later and gave information regarding participation in cardiac rehabilitation during the follow up year.
Measure: Number; unit: events
Units Other Than Participants: hospitalizations
Arm/Group | Education (Intervention) Regarding Cardiac Rehabilitation (CR) | No Education (Control) Regarding Cardiac Rehabilitation (CR)
Number analyzed (Participants) | 413 | 441
Number analyzed (hospitalizations) | 221 | 292
events
  Acute myocardial infarction (MI) | 61 | 84
  Acute, but ill-defined cerebrovascular disease (a | 31 | 35
  Angina Pectoris | 6 | 8

3. Other Pre Specified Outcome: Biochemical Markers
Description: glucose, total cholesterol, triglycerides, low density lipoprotein (LDL) cholesterol. Data regarding these biochemical markers was collected from medical available documents at the homes of the patients. In many cases this data was unavailable. Reported values are only available for a subpopulation.
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Education (Intervention) Regarding Cardiac Rehabilitation (CR) | No Education (Control) Regarding Cardiac Rehabilitation (CR)
Number analyzed (Participants) | 413 | 441
mg/dl
  Glucose | 120.4 (58.0) [115.9 to 124.8] | 123.1 (64.8) [118.3 to 128.0]
  Total Cholesterol | 164.4 (38.5) [160.0 to 168.7] | 170.6 (43.5) [165.8 to 175.4]
  Triglycerides | 141.7 [134.0 to 149.4] | 142.1 [133.6 to 150.6]
  LDL Cholesterol | 95.3 [91.5 to 99.1] | 96.8 [92.8 to 100.8]

4. Other Pre Specified Outcome: Medical Service Utilization
Description: Visits to the emergency department during the year following CABG surgery
Time Frame: 1 year
Measure: Number; unit: ER visits
Arm/Group | Education (Intervention) Regarding Cardiac Rehabilitation (CR) | No Education (Control) Regarding Cardiac Rehabilitation (CR)
Number analyzed (Participants) | 413 | 441
ER visits | 78 | 74

5. Other Pre Specified Outcome: Anthropometric Measures
Description: Measurements of body mass index (BMI)
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Education (Intervention) Regarding Cardiac Rehabilitation (CR) | No Education (Control) Regarding Cardiac Rehabilitation (CR)
Number analyzed (Participants) | 413 | 441
kg/m^2
  Body Mass Index (BMI) men | 28.0 (4.4) [27.6 to 28.4] | 27.3 (4.4) [26.9 to 27.7]
  Body Mass Index (BMI) women | 28.9 [27.9 to 30.0] | 28.4 [27.6 to 29.3]

6. Other Pre Specified Outcome: Lifestyle Habits (i.e. Smoking)
Time Frame: 1 year
Measure: Number; unit: patients
Arm/Group | Education (Intervention) Regarding Cardiac Rehabilitation (CR) | No Education (Control) Regarding Cardiac Rehabilitation (CR)
Number analyzed (Participants) | 413 | 441
patients
  Current smoker | 38 | 46
  Past smoker | 208 | 215
  Never smoked | 157 | 167

7. Other Pre Specified Outcome: Employment Status
Description: Number of patients fully employed in each arm
Time Frame: 1 year
Measure: Number; unit: patients
Arm/Group | Education (Intervention) Regarding Cardiac Rehabilitation (CR) | No Education (Control) Regarding Cardiac Rehabilitation (CR)
Number analyzed (Participants) | 413 | 441
patients | 88 | 82

8. Other Pre Specified Outcome: Depression & Anxiety
Description: Score in the HADS (hospital Anxiety and Depression Scale) screening for anxiety and depression. This is a 14 item scale, 7 items for anxiety and 7 items for depression. Each item can score 0-3 (0=good, 3=bad) and the total score for each scale varies between 0 (no depression/anxiety) to 21 (clinical depression/anxiety requiring medical intervention)
Time Frame: 1 year
Population: All patients who completed the Hospital Anxiety and Depression Scale (HADS)
Measure: Mean (Standard Deviation); unit: HADS score
Arm/Group | Education (Intervention) Regarding Cardiac Rehabilitation (CR) | No Education (Control) Regarding Cardiac Rehabilitation (CR)
Number analyzed (Participants) | 413 | 441
HADS score
  Anxiety (0=low; 21=high) | 4.66 (4.08) | 5.33 (4.21)
  Depression (0=low ; 21=high) | 4.49 (4.32) | 4.66 (4.09)

9. Other Pre Specified Outcome: Physical Activity
Description: Self-reported physical activity using a physical activity questionnaire validated in Hebrew. Details of the study validating the instrument: "Development of a Hebrew questionnaire to be used in epidemiological studies to assess physical fitness--validation against sub maximal stress test and predicted VO2max". Ken-Dror G, Lerman Y, Segev S, Dankner R. Harefuah. 2004 Aug;143(8):566-72, 623. Hebrew. PMID: 15523807 VO2max=maximal oxygen uptake
Time Frame: 1 year
Population: All patients who were interviewed 1-year after CABG surgery and responded to the physical activity questionnaire
Measure: Number; unit: patients
Arm/Group | Education (Intervention) Regarding Cardiac Rehabilitation (CR) | No Education (Control) Regarding Cardiac Rehabilitation (CR)
Number analyzed (Participants) | 413 | 441
patients
  Physically active in any sports | 190 | 162
  Sedentary (no sports activities) | 223 | 279

10. Secondary Outcome: MacNew Heart Disease Health Related Quality of Life (HRQL) Scale. A Self-administered Heart Disease-specific Health-related Quality of Life (HRQL) Instrument.
Description: MacNew questionnaire (MACNEW). A self-administered heart disease-specific health-related quality of life (HRQL) instrument. The MacNew is a modification of the original interviewer-administered Quality of Life after Myocardial Infarction [QLMI] instrument. It addresses three major HRQL domains, the Emotional, Physical, and Social domains which can be combined to give a Global HRQL score. The MacNew consists of 27 items. The total mean score ranges between 1 and 7, where higher score means better HRQL.
Time Frame: 1 year
Population: The N for this outcome is the number of patients for whom there are follow-up data after one year.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Educational (Intervention) on Cardiac Rehabilitation (CR): Cardiac patients were encouraged to participate in cardiac rehabilitation (CR) following coronary artery bypass grafting (CABG) surgery. Medical staff in the operating cardiothoracic units (surgeons and nurses) were encouraged to refer patients to CR.
- No Education (Control) About Cardiac Rehabilitation (CR): Cardiac patients undergoing coronary artery bypass grafting (CABG) surgery receive the usual care without being exposed to the educational intervention. The staff in the cardiothoracic units (surgeons and nurses) did not receive any information about cardiac rehabilitation (CR) and were giving the usual care.
Arm/Group | Educational (Intervention) on Cardiac Rehabilitation (CR) | No Education (Control) About Cardiac Rehabilitation (CR)
Number analyzed (Participants) | 413 | 441
Scores on a scale | 5.58 (0.94) | 5.27 (0.89)

11. Other Pre Specified Outcome: Blood Pressure
Description: The pooled mean of 3 blood pressure measurements taken during the interview
Time Frame: 1 year follow up
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Education (Intervention) Regarding Cardiac Rehabilitation (CR) | No Education (Control) Regarding Cardiac Rehabilitation (CR)
Number analyzed (Participants) | 450 | 454
mm Hg
  Systolic | 131.9 [130.1 to 133.7] | 130.8 [129.1 to 132.5]
  Diastolic | 74.6 [73.8 to 75.5] | 74.6 [73.8 to 75.4]

ADVERSE EVENTS:
Time Frame: 1-year follow up after baseline interview.
Description: Baseline interview was conducted during hospitalization period before CABG surgery.
Arm/Group | Education (Intervention) Regarding Cardiac Rehabilitation (CR) | No Education (Control) Regarding Cardiac Rehabilitation (CR)
Serious Adverse Events (participants affected / at risk) | 114/504 | 159/523
Other Adverse Events (participants affected / at risk) | 0/504 | 0/523
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Education (Intervention) Regarding Cardiac Rehabilitation (CR) (N=504) | No Education (Control) Regarding Cardiac Rehabilitation (CR) (N=523)
Death (Cardiac disorders) | 16 (16) | 32 (32) — Total mortality
acute myocardial infarction, unspecified site (Cardiac disorders) | 61 (61) | 84 (84)
acute, but ill-defined cerebrovascular disease (apoplexy, n.o.s)/transient cerebral ischemia (Vascular disorders) | 31 (31) | 35 (35)
other and unspecified angina pectoris (Cardiac disorders) | 6 (6) | 8 (8)

LIMITATIONS AND CAVEATS:
1. Lack of randomization
2. No biochemical tests were performed by the study and information regarding biochemical parameters was drawn from the medical records during baseline and from medical documents during follow up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes